CLINICAL TRIAL: NCT01151280
Title: A Multi-Center, Prospective Study the WallFlex Biliary RX Fully Covered Stent for the Treatment of Anastomotic Biliary Strictures in Post Liver Transplant Patients.
Brief Title: WallFlex Biliary Post Liver Transplant IDE Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7055; E7055 (Other: Boston Scientific)
Record Dates: First submitted 2010-06-21; First posted 2010-06-28 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Anastomotic Biliary Stricture Post Orthotopic Liver Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WallFlex Biliary Fully Covered Stent (Experimental): All eligible patients entered into the study will be treated with a WallFlex Biliary Fully Covered Stent
  Interventions: Device: WallFlex Biliary Fully Covered Stent

INTERVENTIONS:
Device: WallFlex Biliary Fully Covered Stent — Investigational device evaluated for the treatment for benign biliary strictures

SUMMARY:
The primary objective of this study is to demonstrate effectiveness of the WallFlex Biliary RX Fully Covered Stent for anastomotic biliary strictures in post-orthotopic liver transplant (OLT) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Post -OLT patients with symptoms of biliary obstruction secondary to anastomotic biliary stricture as assessed by:

   * Clinical signs and symptoms including jaundice, abdominal pain, pruritis, and cholangitis
   * Abnormal liver function tests (serum bilirubin > 1.5 and/or elevated alkaline phosphatase levels)
   * Abnormal imaging on ultrasound, CT scan, or MRCP suggestive of a biliary stricture
3. Willingness and ability to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Roux-en-Y choledochojejunostomy
2. Suspected nonanastomotic biliary strictures based on imaging(i.e. multiple strictures, strictures that are longer than 8cm in length, strictures located in the intrahepatic ducts and/or in the donor duct proximal to the site of anastomosis)
3. Living donor transplants
4. Transplants performed within 30 days (fresh transplants)
5. Perforation of any duct within the biliary tree
6. Patients with known sensitivity to any components of the stent or delivery system
7. Patients with malignancy involving the biliary tree (including hepatocellular carcinoma)
8. Patients with poor Karnofsky score
9. Life expectancy of less than one year
10. Inability to pass a guidewire through the strictured area
11. Previous biliary metal or multiple plastic stent placement
12. Drug-induced or cholestatic hepatitis from an infective cause
13. Redundant bile duct that may be treated by temporary placement of stent or conversion to a RouxEnY hepaticojejunostomy
14. Choledocholithiasis/biliary "cast" syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Divyesh Sejpal, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai Medical Center, New York, New York
  - Mansour Parsi, MD, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who signed an informed consent form and met the inclusion/exclusion criteria for this study were enrolled. The first subject was enrolled for this study on October 06, 2009 and the last subject was enrolled on February 01, 2012.
Groups:
- WallFlex Biliary Fully Covered Stent: Patients who signed an informed consent form and who met the inclusion/exclusion criteria for the study received a WallFlex Biliary Fully Covered Stent for treatment of anastomotic stricture post orthotopic liver transplant.
Period: Overall Study
Arm/Group | WallFlex Biliary Fully Covered Stent
Started | 10
Completed | 6
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: All participants were included for analysis.
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (5.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Stricture Resolution at the Time of Stent Removal.
Description: Stricture resolution is assessed at the time of stent removal. Stricture resolution is confirmed by cholangiogram and/or balloon sweep of the biliary duct. Stent removal can be per-protocol (3 months indwell) or early.
Time Frame: At 3 months (per protocol removal) or at early removal.
Population: All participants were included for analysis.
Measure: Number; unit: participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 10
participants
  Participants with resolution at removal | 9
  Participants without resolution at removal | 1

2. Secondary Outcome: Safety
Description: Safety is being measured by the occurrence, severity, device- and procedure-relatedness of adverse events during stent placement, during stent indwell, at the time of stent removal, and after stent removal.
  Unit of measure will be the actual number of adverse events that occurred.
Time Frame: From enrollment through end of study.
Population: All participants were included for analysis.
Measure: Number; unit: adverse events
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 10
adverse events
  Device Related Adverse Event | 2
  Placement Procedure Related Adverse Event | 2
  Removal Procedure Related Adverse Events | 0

3. Secondary Outcome: Stent Removability
Description: Stent removability is measured as the ability to successfully remove the stent at initial placement in case of inadequate stent placement, during the stent indwell period in case of stent failure, or at the end of indwell without any clinically significant complications or technical difficulties. A clinically significant complication is defined as a medical event that requires an intervention.
Time Frame: At 3 months (per protocol removal) or early removal
Population: All participants were included for analysis.
Measure: Number; unit: participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 10
participants
  Successful Removal | 9
  Stent not removed due to migration out of duct | 1

4. Secondary Outcome: Technical Success of Stent Placement
Description: Evaluation of technical success of the stent placement defined as the ability to deploy the stent in satisfactory position across the stricture as determined by cholangiogram.
Time Frame: At stent placement (Day 1)
Population: All participants were included for analysis.
Measure: Number; unit: participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 10
participants
  Technical Success Achieved | 10
  Technical Success Not Achieved | 0

5. Secondary Outcome: Effectiveness of Stent at 6 Months
Description: Evaluation of effectiveness of the stent by assessing for resolution of stricture at 6 months as determined by cholangiogram.
  "Effectiveness" is defined as the absence of biliary obstructive symptoms after receiving a WallFlex stent.
  Subjects received liver function tests at the 1 Month and 6 Month post stent removal follow-up visits and were also assessed for biliary obstructive symptoms.
Time Frame: From stent removal through 6 months post stent removal follow-up.
Population: Effectiveness was assessed in 9 participants that had stricture resolution at the time of stent removal. 1 participant did not have resolution at removal and therefore could not be assessed in the post stent removal follow-up period.
Measure: Number; unit: participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 9
participants
  Maintained Resolution 6 Months Post Removal | 6
  Recurrence of Biliary Stricture | 2
  Discontinued due to Unrelated Adverse Event | 1

6. Secondary Outcome: Re-intervention Occurrence
Description: Evaluation of the occurrence of re-intervention. Re-intervention is defined as any type of endoscopic, percutaneous, or surgical procedure to improve biliary drainage during stent indwell or through 6 months of follow-up after stent removal.
Time Frame: 6 months post stent removal
Population: All participants were included for analysis.
Measure: Number; unit: participants
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 10
participants
  No Reintervention | 4
  Endoscopic Reintervention - Stent Removed | 2
  Endoscopic Reintervention - Re-stented | 2
  Endo Reintervention - Stent Removed and Re-stented | 1
  Percutaneous Reintervention - Drainage | 1

7. Secondary Outcome: Time to Stent Occlusion
Description: Evidence of stent occlusion
  "stent occlusion" was assessed during the stent indwell period (from stent placement procedure through the stent removal procedure. 3 months according to protocol). Subjects received liver function tests at the 48 hour, Week 1, Month 1, and Month 3 stent indwell follow-up visits and were also asked if they were experiencing biliary obstructive symptoms at each visit. If stent occlusion was suspected, imaging and/or endoscopic intervention was performed. One subject experienced stent occlusion at 68 days post stent placement. Time to event data was not generated as not enough events occurred to calculate medial time to event data.
Time Frame: mean time from stent placement to stent removal for all 10 patients was 91.3 days.
Population: All participants were included for analysis.
  1/10 subjects experienced stent occlusion at 68 days post stent placement. Mean time to event data was not calculated as only 1 stent occlusion occurred in 10 subjects.
Measure: Number; unit: days
Arm/Group | WallFlex Biliary Fully Covered Stent
Number analyzed (Participants) | 10
days | 68

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all participants from the time of informed consent through the final follow-up visit.
Arm/Group | WallFlex Biliary Fully Covered Stent
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WallFlex Biliary Fully Covered Stent (N=10)
General abdominal pain (Hepatobiliary disorders) | 1 (1) — Related to stent placement procedure
Post-ERCP (endoscopic retrograde cholangiopancreatography) pancreatitis (Hepatobiliary disorders) | 1 (1) — Related to stent placement procedure
Elevated bilirubin (Hepatobiliary disorders) | 1 (1) — Related to device
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Recurrence of biliary stricture (Hepatobiliary disorders) | 2 (2) — Recurrence of biliary stricture was an adverse event that occurred in 2 participants. Both adverse events were unrelated.
Altered mental status (Hepatobiliary disorders) | 1 (1) — Unrelated
Hyponatremia (Blood and lymphatic system disorders) | 1 (1) — Unrelated
Cholangitis (Hepatobiliary disorders) | 1 (1) — Unrelated
Hepatic artery thrombosis (Vascular disorders) | 1 (1) — Unrelated
Acute renal failure (Renal and urinary disorders) | 1 (1) — Unrelated
Anemia (Metabolism and nutrition disorders) | 1 (1) — Unrelated
Pulmonary vascular congestion (Vascular disorders) | 1 (1) — Unrelated
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1) — Unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WallFlex Biliary Fully Covered Stent (N=10)
Right upper quadrant pain (Hepatobiliary disorders) | 2 (2) — This AE occurred in 2 participants. One occurrence was related to the device The second occurrence was unrelated
Dark urine (Hepatobiliary disorders) | 1 (1) — Unrelated
Pale stools (Hepatobiliary disorders) | 1 (1) — Unrelated
Itching (Hepatobiliary disorders) | 3 (3) — This AE occurred in 3 participants. All 3 occurrences were unrelated

LIMITATIONS AND CAVEATS:
This was a small, pilot, feasibility study. Further prospective studies are needed to optimize duration of fully covered self-expanding metal stent indwell and assess predictors of treatment success.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No